CLINICAL TRIAL: NCT01213849
Title: An Open-label, Randomised, 3-way Crossover Single Dose Study to Demonstrate Dose Proportionality of Fluticasone Furoate (FF) and Equivalence of Vilanterol (VI) When Administered as FF/VI Inhalation Powder From the Novel Dry Powder Inhaler in Healthy Subjects.
Brief Title: Dose Proportionality Study: Blood Levels of Fluticasone Furoate (FF) and Vilanterol (VI) Following Different Doses of FF/VI Via an Inhaler
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 102932
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 200/100 mcg fluticasone furoate/vilanterol (Experimental): 4 inhalations of 50/25 mcg fluticasone furoate/vilanterol
  Interventions: Drug: Fluticasone furoate 50 mcg (4 inhalations); Drug: Vilanterol 25 mcg (4 inhalations)
- 400/100 mcg fluticasone furoate/vilanterol (Experimental): 4 inhalations of 100/25 mcg fluticasone furoate/vilanterol
  Interventions: Drug: Fluticasone furoate 100 mcg (4 inhalations); Drug: Vilanterol 25 mcg (4 inhalations)
- 800/100 mcg fluticasone furoate/vilanterol (Experimental): 4 inhalations of 200/25 mcg fluticasone furoate/vilanterol
  Interventions: Drug: Fluticasone furoate 200 mcg (4 inhalations)

INTERVENTIONS:
Drug: Fluticasone furoate 50 mcg (4 inhalations) — 4 inhalations of 50 mcg strength
  Arms: 200/100 mcg fluticasone furoate/vilanterol
Drug: Fluticasone furoate 100 mcg (4 inhalations) — 4 inhalations of 100 mcg strength
  Arms: 400/100 mcg fluticasone furoate/vilanterol
Drug: Fluticasone furoate 200 mcg (4 inhalations) — 4 inhalations of 200 mcg strength
  Arms: 800/100 mcg fluticasone furoate/vilanterol
Drug: Vilanterol 25 mcg (4 inhalations) — 4 inhalations of 25 mcg strength
  Arms: 200/100 mcg fluticasone furoate/vilanterol; 400/100 mcg fluticasone furoate/vilanterol

SUMMARY:
The purpose of this study is to demonstrate dose proportionality of fluticasone furoate (FF) and equivalence of vilanterol (VI)following single dose administration of FF/VI via the novel dry powder inhaler in healthy subjects.

DETAILED DESCRIPTION:
The study will be an open-label, randomised, 3-way cross-over single dose study in 24 healthy subjects to demonstrate dose proportionality of fluticasone furoate (FF) and equivalence of vilanterol (VI) following single dose administration of FF/VI via the novel dry powder inhaler. In each of 3 treatment periods, subjects will receive 4 inhalations of 50/25 mcg, 100/25 mcg, 200/25 mcg FF/VI. Blood samples will be taken for pharmacokinetic analysis and safety (12-lead ECGs, clinical laboratory test, vital signs, adverse events) will be monitored following each dose.

ELIGIBILITY:
Inclusion Criteria:

* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <or= 1.5xULN
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age inclusive.
* A female subject is eligible to participate if she is of:

Non-child-bearing potential defined as post-menopausal females with a documented tubal ligation or hysterectomy, or postmenopausal defined as 12 months of spontaneous amenorrhea.

Child-bearing potential and agrees to use one of the approved contraception methods until 16 weeks after the last dose.

* Male subjects with female partners of child-bearing potential must agree to use one of the approved contraception methods until 16 weeks after the last dose.
* Body Mass Index (BMI) within range 18.5-29.0 kg/m2 (inclusive).
* Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcF < 450 msec.
* No clinically significant abnormality on the Holter electrocardiogram (ECG) at screening.
* Subjects who are current non-smokers, who have not used any tobacco products in the 12 month period preceding the screening visit, and have a pack history of < or = 5 pack years.
* Able to satisfactorily use the dry powder inhaler.

Exclusion Criteria:

* As a result of medical interview, physical examination or screening investigations, the principal investigator or delegate physician deems the subject unsuitable for the study. Subjects must not have a systolic blood pressure above 145 mmHg or a diastolic pressure above 85 mmHg unless the Investigator confirms that it is satisfactory for their age.
* The subject has a history of breathing problems in adult life (e.g. history of asthmatic symptomatology). Screening lung function tests (forced expiratory volume in 1 minute (FEV1)) will be performed to confirm normal lung function parameters (>or=85% predicted).
* Subjects who have suffered a lower respiratory tract infection within 4 weeks of the screening visit.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
* A positive HIV antibody.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* History of heavy regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females.
* History or regular use of tobacco- or nicotine-containing products within 12 months prior to screening.
* Positive carbon monoxide or alcohol breath test at screening or on admission to the unit.
* A positive pre-study urine drug screen or when randomly tested during the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has taken systemic, oral or depot corticosteroids less than 12 weeks before the screening visit.
* The subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
* History of sensitivity or adverse reaction to any of the study medications including immediate or delayed hypersensitivity to any beta-agonist, sympathomimetic drug, or an intranasal, inhaled or systemic corticosteroid; known suspected sensitivity to the constituents of the new powder inhaler (lactose or magnesium stearate) or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates participation.
* History of severe milk protein allergy.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months of the start of the study.
* Pregnant females as determined by positive serum hCG test at screening or by positive serum/urine hCG test prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10-04 (Actual); Primary Completion 2010-11-25 (Actual); Study Completion 2010-11-25 (Actual)

PRIMARY OUTCOMES:
Fluticasone furoate area under concentration-time curve (AUC) | 48 hours post-dose
Fluticasone furoate maximum observed concentration (Cmax) | 48 hours post-dose
Vilanterol area under concentration-time curve (AUC) | 48 hours post-dose
Vilanterol maximum observed concentration (Cmax) | 48 hours post-dose

SECONDARY OUTCOMES:
Fluticasone furoate time of occurence of maximum concentration (tmax) | 48 hours post-dose
Vilanterol time of occurence of maximum concentration (tmax) | 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 102932 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/102932?search=study&search_terms=102932#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 102932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 102932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 102932 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register